CLINICAL TRIAL: NCT07054502
Title: Prospective Validation of Deep Learning Model to Predict Postoperative Major Adverse Cardiac and Cerebrovascular Event
Brief Title: Prospective Validation of DL Model for Postoperative MACCE Prediction
Status: Not yet recruiting | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hyun-Kyu Yoon, Clinical Associate Professor, Seoul National University Hospital
Other Study IDs: 2503-210-1630
Record Dates: First submitted 2025-06-27; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Major Adverse Cardiovascular and Cerebrovascular Events (MACCE)
Keywords: Deep learning; Non-cardiac surgery; Electrocardiogram; Multimodal; MACCE

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Non-cardiac surgical patients: Patient undergoing non-cardiac surgery under regional or general anesthesia

SUMMARY:
This study aims to prospectively validate a deep learning model developed using retrospective data to predict major adverse cardiac and cerebrovascular events (MACCE) occurring within 30 days after non-cardiac surgery. The validation will be performed using prospectively collected data from patients undergoing non-cardiac surgery under general or regional anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 or older undergoing non-cardiac surgery under general or regional anesthesia at Seoul National University Hospital

Exclusion Criteria:

* Reoperation within 30 days after initial surgery
* Organ procurement or pregnancy-related procedures
* Ambulatory-based surgery
* Preoperative tracheal intubation before entering the operating room
* Surgeries performed outside the operating room

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non-cardiac surgical patients
Sampling Method: Non-Probability Sample
Enrollment: 7000 (Estimated)
Dates: Start 2025-07-10 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiovascular and cerebrovascular events (MACCE) | within 30 days after surgery
  Occurrence of MACCE within 30 days after surgery (composite outcome including myocardial infarction, stroke, coronary revascularization, heart failure, and death)

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No